CLINICAL TRIAL: NCT05474742
Title: The Nori Health App: (Pilot) Randomized Controlled Trial
Brief Title: The Nori Health App
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: bankruptcy app owner
Sponsor: UMC Utrecht (Other)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Elke Mathijssen, Principal investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nori_Health
Record Dates: First submitted 2022-07-08; First posted 2022-07-26 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: IBD; Crohn Disease; Ulcerative Colitis
Keywords: Randomized Controlled Trial; Pilot; Qualitative component
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Use of the Nori Health app during the study period, standard care
  Interventions: Other: The Nori Health app
- Control group (No Intervention): No use of the Nori Health app during the study period, standard care

INTERVENTIONS:
Other: The Nori Health app — The Nori Health app consist of a chatbot that instantly answers questions about topics relevant to patients with IBD and 6-week education program. The chatbot is driven by artificial intelligence and armed with state of the art scientific literature to offer to the right information to the right person at the right time. The education program is offered during the first six weeks of use. The Nori Health app then actively offers information on four fixed topics and two topics to a participant's choosing (i.e. low energy, pain, stress, mental health, hydration, exercising). It is expected from participants that they respond to this by having approximately five chat conversations of five minutes per week. Participants in the intervention group receive access to the Nori Health app for a 6-month period directly after randomization. They are free to use the Nori Health app whenever and as often as they want. Participants in the control group receive no intervention.
  Arms: Intervention group

SUMMARY:
A multicenter, randomized controlled trial with an embedded pilot and qualitative component to investigate the effects of the Nori Health app.

DETAILED DESCRIPTION:
RATIONALE Inflammatory bowel disease (IBD) is an umbrella term used to describe diseases that involve chronic inflammation of the gastrointestinal tract. Although progress in treatment has been made over the past two decades, IBD continues to profoundly affect patients' quality of life. Since patients with IBD have to deal with their disease's complex and unpredictable nature 24 hours a day, it is important that they have access to self-management support outside the hospital. Nori Health aims to provide this support with an app that consists of an artificial intelligence-driven chatbot and 6-week education program.

OBJECTIVES

The primary objective is to investigate whether use of the Nori Health app improves the level of patient activation for self-management in patients with IBD by comparing an intervention and (waiting-list) control group at 6 weeks after randomization. Secondary objectives are:

* To investigate whether there are any differences between the intervention and control group in the level of patient activation for self-management at 12 and 20 weeks after randomization;
* To investigate whether there are any differences between the intervention and control group in the level of disease control at 6, 12 and 20 weeks after randomization;
* To investigate whether there are any differences between the intervention and control group in quality of life at 6, 12 and 20 weeks after randomization;
* To investigate whether there are any differences between the intervention and control group in healthcare utilization at 6, 12 and 20 weeks after randomization;
* To investigate intervention fidelity at 6, 12 and 20 weeks after randomization;
* To explore the experiences of patients with IBD with use of the Nori Health app and their views on its pros and cons.

STUDY DESIGN A multicenter, randomized controlled trial with an embedded pilot and qualitative component.

STUDY POPULATION

Patients with IBD are eligible for participation if they:

* Are aged >18 years;
* Are able to read and write the Dutch language;
* Are in the possession of a tablet or smartphone with WiFi connection.

Excluded are those with cognitive impairments or who are already familiar with use of the Nori Health app.

STUDY INTERVENTION Participants are randomized in a 1:1 ratio to the intervention or control group. Participants in the intervention group receive access to the Nori Health app for a 6-month period directly after randomization. They are free to use the Nori Health app whenever and as often as they want. Participants in the control group receive no intervention. Standard IBD care continues unchanged. After study completion, participants in the control group also receive access to the Nori Health app for a 6-month period.

STUDY PARAMETERS The level of patient activation for self-management is assessed using the patient activation measure. The IBD control questionnaire and EQ-5D are used to assess respectively the level of disease control and quality of life. Healthcare utilization is assessed with 5 close-ended questions. System data is used to assess intervention fidelity. Experiences of patients with IBD with use of the Nori Health app and their views on its pros and cons are explored by performing individual, semi-structured, telephonic interviews.

ELIGIBILITY:
Patients with IBD are eligible for participation if they:

* Are aged >18 years;
* Are able to read and write the Dutch language;
* Are in the possession of a tablet or smartphone with WiFi connection.

Excluded are those with cognitive impairments or who are already familiar with use of the Nori Health app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | 6 weeks follow-up
  Measure of patient activation for self-management. Scale from 0 to 100, higher scores mean a higher level of patient activation for self-management (=better outcome).

SECONDARY OUTCOMES:
Patient Activation Measure (PAM) | 12 and 20 weeks follow-up
  Measure of patient activation for self-management. Scale from 0 to 100, higher scores mean a higher level of patient activation for self-management (=better outcome).
Inflammatory Bowel Disease (IBD)-control questionnaire | 6, 12 and 20 weeks follow-up
  Measure of disease control. Scale from 0 to 16, higher scores mean a higher level of disease control (=better outcome).
EuroQol-5 dimension questionnaire (EQ-5D) | 6, 12 and 20 weeks follow-up
  Measure of quality of life. Scale from 0 to 100, higher scores mean a higher quality of life (=better outcome).
Healthcare utilization | 6, 12 and 20 weeks follow-up
  Brief questionnaire with 5 close-ended questions on healthcare utilizatio, using a nominal scale (e.g., yes/no).

OTHER OUTCOMES:
Interviews | 6-20 weeks follow-up
  Experiences of patients with IBD with use of the Nori Health app and their views on its pros and cons.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391